CLINICAL TRIAL: NCT04928937
Title: Pharmacokinetics of SSRI/SNRI (Selective Serotonin Reuptake Inhibitors/ Serotonin-norepinephrine Reuptake Inhibitors) After Bariatric Surgery and the Effects on Clinical Course
Brief Title: Pharmacokinetics of SSRI/SNRI After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: University Hospital, Zürich (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2021IJO00233
Record Dates: First submitted 2021-06-03; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Depression
Keywords: SSRI/SNRI; bariatric surgery
MeSH Terms: conditions — Obesity; Depression | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bariatric surgery: consisting of gastric bypass surgery: Roux-en-Y gastric bypass (RYGB), sleeve gastrectomy (SG)
  Interventions: Procedure: Roux-en-Y gastric bypass, sleeve gastrectomy
- conservative therapy: consisting of medical visits, nutritional counseling, physiotherapy, anti-obesogenic medication and psychological coaching

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass, sleeve gastrectomy — bariatric surgery with the goal loosing weight
  Groups: bariatric surgery

SUMMARY:
Psychiatric disorders and treatment with antidepressants SSRI/SNRI (selective serotonin reuptake inhibitors/ serotonin-norepinephrine reuptake inhibitors) are common in people with morbid obesity who are candidates for bariatric surgery. Although longitudinal assessments reveal positive effects of bariatric surgery on quality of life and mood, depressive disorders may also deteriorate after bariatric surgery. There is few and inconsistent data about the postoperative pharmacokinetics of SSRI/SNRI. The aims of our study were to provide comprehensive data about the postoperative bioavailability of SSRI/SNRI, and the clinical effects on the course of depression.

DETAILED DESCRIPTION:
Prospective multicenter study including 63 patients (i.e. 46 participants in the bariatric surgery group, and 17 participants in the conservative group as controls) with morbid obesity and therapy with SSRI/SNRI: participants filled the Beck Depression Inventory II (BDI) questionnaire, and plasma levels of SSRI/SNRI were measured by HPLC (High Performance Liquid Chromatography), preoperatively (T0), 4 weeks (T1) and 6 months (T2) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* BMI >35
* Existing antidepressant drug therapy with SSRI or SNRI
* Written informed consent

Exclusion Criteria:

* Taking other psychotropic drugs than SSRI/SNRI
* Active drug addiction or psychosis
* Severe depression (BDI score >30)
* Suicidality at the beginning of the study
* Gastrointestinal malabsorption
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As part of the regular consultation at the obesity center of the three study sites patients were assessed for participation according to the inclusion and exclusion criteria of the study. An interprofessional team decided about the treatment, consisting of gastric bypass surgery (Roux-en-Y gastric bypass [RYGB]), sleeve gastrectomy (SG) or conservative therapy (consisting of medical visits, nutritional counseling, physiotherapy, antiobesogenic medication and psychological coaching). Afterwards, patients who had met the inclusion criteria were asked for participation, and were allocated (according to the treatment option) to the "bariatric surgery group" with the two subgroups "gastric bypass" and "sleeve gastrectomy", and to the "conservative group".
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in SSRI/SNRI blood levels after surgery | Change in SSRI/SNRI blood levels at 4 weeks and 6 months after surgery
  Blood analysis: blood samples were drawn at the predefined time period (corresponding to the presumed Tmax) after ingesting the SSRI/SNRI
Change in BDI (Beck Depression Inventory) II questionnaire scores after surgery | Change in BDI II questionnaire scores at 4 weeks and 6 months after surgery
  The BDI is a psychological test that measures the severity of depressive symptoms or depression. The test procedure is a self-assessment measure including 21 questions on a four-level scale with values from 0 to 3 in terms of occurrence and intensity, providing a sum value between 0 and 63. Based on this value, it is possible to determine whether the person is non-depressed (0), minimally depressed, mildly depressed, moderate to severely depressed or severely depressed (63).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pasi, MD, Principal Investigator — Universitätsspital Zürich
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No